CLINICAL TRIAL: NCT05662839
Title: Feasibility of Utilising Brushing Cytology and Dermoscopy for Diagnosing Penile Lesions
Acronym: BRUCY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CFTSp203
Record Dates: First submitted 2022-10-03; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Penile Cancer
Keywords: Penile cancer; HPV; Cytology testing
MeSH Terms: conditions — Penile Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to one of two groups. Each group will receive standard of care and the additional procedures being investigated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research Arm (Experimental): Each group will undergo the same study procedures; Dermoscope Cytological brushing Complete questionnaire on experience of the cytological brushing SoC treatment
  Interventions: Device: Cytological Brushing

INTERVENTIONS:
Device: Cytological Brushing — All participants will undergo cytological brushing to collect cell samples for analysis

SUMMARY:
In an attempt to reduce patient flow into the hospital we are going to assess the use of penile cytological brushings and dermoscopy in diagnosing cancer or non-cancer conditions of the penis.

DETAILED DESCRIPTION:
Currently the standard of care pathway for all patients suspected of having penile cancer involves the need for a penile biopsy under local (LA) or general anaesthetic (GA). We hope to assess the feasibility of cytololgical brushings and the patient experience of the use of such a technique. Additionally, we will make initial comparison on the concordance between cytological brushing and dermoscope photo vs actual biopsy only.

Importantly for this study, all patients will be offered standard of care: a biopsy under LA or GA. The additional procedures of the cytological brushing and dermoscope photo will be done in an out-patient clinic setting (with no anaesthetic).

If it can be shown that the inclusion of the cytological brushing and dermoscope photo have comparative results over current standard of care histological biopsy, this will provide sufficient evidence to expand this study to acquire more data.

ELIGIBILITY:
Inclusion Criteria:

1. All patients requiring either diagnostic biopsy or WLE (wide local excision) of a lesion of the penis
2. Age > 18 years
3. Written informed consent provided by the patient
4. Subject has been scheduled for surgical intervention, with a biopsy procedure being a part of the surgical plan

Exclusion Criteria:

1. Subject is unfit for surgery upon surgeon's assessment.
2. Unable to provide consent
3. Those with terminal disease
4. Those with palpable lymph nodes
5. Other coincident cancers
6. Previous radiotherapy treatment to the penis, bladder, prostate, anus
7. Subject is deprived of liberty or under guardianship
8. Subject is not able to follow and understand the procedures of the study due to mental state or other reasons

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Does cytology results compare equally with standard histological biopsy for detecting cancer | Through study completion, expected to be 12 months
  Concordance of cytology vs Histopathology i.e. is the cytology assessment equal to histopathology results when detecting cancer
Does the use of dermoscopy photography enable us to identify abnormal cellular changes that compare equally to the results obtained with standard histological biopsy. | Through study completion, expected to be 12 months
  Concordance of dermoscopy vs Histopathology in detecting cancer i.e. does the use of dermoscopy photographs enable us to identify cancer and compare equally to results obtained by histopathology

SECONDARY OUTCOMES:
Patient satisfaction with cytological brushing diagnostic method being tested | Through study completion, expected to be 12 months
  All patients on study will be asked their views on the cytology brushing technique being used to gauge their satisfaction and experience of the new diagnostic method being tested

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Sangar, Principal Investigator — The Christie NHS FT

IPD SHARING:
Plan to Share IPD: No
no intention to share individual participant data with other researchers outside of the BRUCY research study.